CLINICAL TRIAL: NCT00657800
Title: The Effect of a Coordinated Inpatient Diabetes Education Program on Glycemic Control, Diabetes Self-Management, Patient Satisfaction, and Quality of Life in the Outpatient Setting
Brief Title: The Effect of a Coordinated Inpatient Diabetes Education Program in the Outpatient Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Mary T. Korytkowski, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PRO07030238
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2010-09-22 (Estimated); Status verified 2010-09

CONDITIONS: Diabetes
Keywords: diabetes, inpatient, education,
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Behavioral - Intensified coordinated inpatient diabetes education program (IDEP)
  Interventions: Behavioral: Intensified inpatient diabetes education program (IDEP)
- Group 2 (No Intervention): Diabetes education as is typically provided by clinical staff

INTERVENTIONS:
Behavioral: Intensified inpatient diabetes education program (IDEP) — Assessment of educational needs and coordination of inpatient unit based education program by Certified Diabetes Educator (CDE)
  Arms: Group 1

SUMMARY:
Patients will be recruited from comparable inpatient units that have been randomized as either interventional (Group 1) or control (Group 2) units. Patients in the interventional group will receive a comprehensive individualized diabetes education program coordinated by a certified diabetes educator. Patients in Group 2 will receive education from clinical staff as it is typically provided. Assessment of patient satisfaction with both inpatient and outpatient care, quality of life, and diabetes self-management skills (including emergency room visits and readmissions) will be measured using surveys completed during hospitalization and 4 months after discharge to determine any differences between the two groups.

DETAILED DESCRIPTION:
Patients will be recruited from matched sets of inpatient units determined to be comparable in terms of staffing and types of patients admitted. One unit from each matched set will be selected as the intervention unit (Group 1) or the control unit (Group 2) as determined by a random draw.

Group 1 patients will receive the coordinated inpatient diabetes education program (IDEP). Patients will be initially evaluated by a certified diabetes educator (CDE) to assess diabetes knowledge and to set priorities for "survival skills" education. Based on this individualized evaluation, a structured education plan will be devised and implemented by the CDE. The structured education plan will be modified as needed throughout the hospital stay to utilize more appropriate educational methods based on patient availability, condition or educational needs.

Group 2 (Control) will receive diabetes education as it is presently provided in our facility by the clinical staff. The staff nurse will be alerted that the patient is a participant in the research study and will record education provided in the electronic medical records.

The modified Michigan Diabetes Research and Training Center's Brief Diabetes Knowledge Test (DKT) and the Diabetes Treatment Satisfaction Questionnaire (DTSQs), if diabetes was pre-existing, will be administered initially to all patients by a member of the research team. If appropriate, the patient will be asked by the research team to complete a Quality of Life Survey (The Medical Outcomes Survey (MOS) Short-Form 36 (SF-36) General Health Survey prior to discharge. Completion of the Diabetes Treatment Satisfaction Questionnaire - Inpatient (DTSQ-IP) will also be requested of the patient prior to discharge.

All participants will be contacted 4 months after discharge for a similar assessment of quality of life and patient satisfaction with diabetes treatment, and for an additional assessment of diabetes self-management practices which includes the number of emergency room visits and readmissions since discharge. Comparisons will be made between the two groups and between baseline and follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with diabetes as defined by ADA criteria
* Ability to understand informed consent document
* Community-dwelling adults

Exclusion Criteria:

* Patients using CSII (continuous subcutaneous insulin infusion)
* Patients with Do Not Resuscitate (DNR) orders
* Decisionally impaired patients
* Patients admitted for 24 hour observation
* Patients in Intensive Care settings
* Patients with language barriers or sensory deficits mandating the need for specialized instruction
* Patients who are pregnant
* Patients for whom transfer to a skilled nursing or other assisted care living facilities is anticipated after discharge.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-12; Primary Completion 2009-10 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Diabetes Self-Management Practices | 4 months post-discharge
Patient Satisfaction | Discharge date, 4 months post-discharge
Quality of Life (QoL) | Baseline and 4 months post-discharge

SECONDARY OUTCOMES:
Glycemic and Metabolic Control | 4 months post-discharge
Emergency Room visits; admissions | 4 months post-discharge

CONTACTS AND LOCATIONS:
Overall Officials: Mary T. Korytkowski, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Department of Medicine, Pittsburgh, Pennsylvania, United States